CLINICAL TRIAL: NCT02574767
Title: Effectiveness on Maternal and Offspring Metabolic Control of a Home-based Dietary and Physical Activity Counseling and n3-long Chain Polyunsaturated Fatty Acids (PUFA) Supplementation in Obese Pregnant Women.
Brief Title: Diet and Physical Activity Counseling and n3-long Chain (PUFA) Supplementation in Obese Pregnant Women
Acronym: MIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); DSM Nutritional Products, Inc. (Industry); Corporación de Apoyo de la Investigación Científica en Nutrición (Other)
Responsible Party: Principal Investigator, Marí-a Luisa Garmendia, Assistant professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fondecyt #1150878
Record Dates: First submitted 2015-10-07; First posted 2015-10-14 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2015-10

CONDITIONS: Obesity; Pregnancy
Keywords: Weight gain, Fatty Acids, Omega-3
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lifestyle counseling + PUFA supplement (Experimental): Home-based Diet and Physical activity plus n3LC-PUFAs supplementation
  Interventions: Behavioral: Lifestyle counseling; Dietary Supplement: PUFA Supplementation
- Routine diet & PA + PUFA Supplementation (Experimental): Routine Diet & Physical Activity counseling care plus n3LC-PUFAs supplementation.
  Interventions: Dietary Supplement: PUFA Supplementation; Behavioral: Routine diet & PA
- Lifestyle counseling + PUFA placebo (Experimental): Home-based Diet and Physical Activity plus placebo for n3LC-PUFAs supplementation.
  Interventions: Behavioral: Lifestyle counseling; Dietary Supplement: PUFA placebo
- Routine diet & PA + PUFA placebo (Placebo Comparator): Routine Diet & Physical Activity counseling plus placebo for n3LC-PUFAs supplementation.
  Interventions: Behavioral: Routine diet & PA; Dietary Supplement: PUFA placebo

INTERVENTIONS:
Behavioral: Lifestyle counseling — Obese pregnant women from PHCC randomized to this group will receive Home-based Diet & Physical activity (PA) counseling. Home-based intervention will consider 2 home visits of one hour of duration. During this session dietary educational and behavioral will be discussed with the participants and their families tailoring the contents based on the specific contexts.
  Arms: Lifestyle counseling + PUFA placebo; Lifestyle counseling + PUFA supplement
Dietary Supplement: PUFA Supplementation — Obese pregnant women from PHCC randomized to this group will receive n3LC-PUFAs oral supplementation based on Schizochytrium oil (S-oil) containing 800 mg docosahexaenoic (DHA) acid/day, which will be administered as capsular preparations containing 200 mg DHA/capsule (4 capsules/day).
  Arms: Lifestyle counseling + PUFA supplement; Routine diet & PA + PUFA Supplementation
Behavioral: Routine diet & PA — Obese pregnant women from PHCC randomized to this group will receive will receive routine diet & PA counseling (i.e. they will receive the standard education sessions included in the prenatal controls at PHCC but no home-based counseling sessions).
  Arms: Routine diet & PA + PUFA Supplementation; Routine diet & PA + PUFA placebo
Dietary Supplement: PUFA placebo — Obese pregnant women from PHCC randomized to this group will receive capsular preparations containing 50 mg DHA/capsule (4 capsules/day), given that evidence suggests that it would be unethical not to provide DHA during pregnancy. Placebo will be delivered in the same way that the n3LC-PUFA supplementation.
  Arms: Lifestyle counseling + PUFA placebo; Routine diet & PA + PUFA placebo

SUMMARY:
In Chile, 1 out of 4 pregnant women is obese (BMI > 30 kg/m2). This impacts negatively the health of the mother and the offspring during pregnancy. Lifestyle interventions are the primary prevention strategy for gestational diabetes in obese women; however, these interventions have shown null or limited effectiveness. In animals, n-3 long-chain polyunsaturated fatty acid (n3LC-PUFAs) have shown to increase insulin sensitivity through higher production and secretion of adipokines, enhanced fatty acids oxidation, reduction of lipogenesis, and direct anti-inflammatory effects; however evidence in humans and during pregnancy is still very limited. Combining a lifestyle intervention with n3LC-PUFAs supplementation could enhance the metabolic control of obese pregnant women. Objective: to assess the effectiveness of two prenatal nutritional interventions (home-based diet and physical activity counseling and/or n3LC-PUFAs supplementation) delivered to obese pregnant women in achieving better metabolic control in both the mother (lower incidence of gestational diabetes mellitus) and the offspring (lower incidence of macrosomia and lower prevalence of insulin resistance at birth).

Methods: this study is a cluster-randomized trial in which obese pregnant women from 12 primary health care centers (PHCC) will be stratified by socio-economic status (SES) and randomized to one of four parallel study arms. We will recruit 1000 women allocated to: 1 Home-based Diet and physical activity (PA) plus n3LC-PUFAs supplementation (Intervention Group 1, n=250); 2. Routine diet & PA counseling care plus n3LC-PUFAs supplementation (Intervention Group 2, n=250); 3. Home-based Diet and Physical activity plus placebo for n3LC-PUFA supplementation (Intervention Group 3, n=250); 4. Routine diet & PA counseling plus placebo (Control Group, n=250). Expected results: we expect that the intervention will contribute to achieving a better metabolic control during pregnancy. Ultimately, we expect that this study will contribute to advance the understanding of how to develop and implement effective actions to promote healthier pregnancies and therefore, healthier lives for mothers and their offsprings.

DETAILED DESCRIPTION:
Obesity and related non-communicable chronic diseases (NCDs: cardiovascular diseases, cancer and diabetes) represent the main causes of death and disability in Chile as well as worldwide. They account for an important proportion of health-care costs and loss of productivity, overloading a country's economy, particularly in developing countries. From a population perspective, it is now clear that preventing the emergence of these conditions is the most effective approach; however most of the current policies fail to incorporate scientific knowledge and thus, are not effective or sustainable. There is now compelling evidence that although obesity and NCDs are mainly observed in adulthood, the risk for most of these conditions originates in the first 1000-days of life (i.e. from pregnancy to two years old). Maternal lifestyle and conditions during pregnancy (e.g. maternal obesity) could affect not only future maternal health, but also risk for NCDs in the next generation. Therefore, pregnancy is a critical window in the implementation of NCDs prevention strategies. Most of the interventions on diet and physical activity (PA) during pregnancy have focused on decreasing gestational weight gain (GWG). Recent meta-analyses of interventions have demonstrated that lifestyle interventions during pregnancy can have a positive effect on GWG. Beyond lifestyle interventions, other dietary interventions have been proposed such as probiotics, vitamin D or n-3 long chain polyunsaturated fatty acids (n3LC-PUFAs) supplementation. Regarding n3LC-PUFAs, differences in plasma fatty acid profiles between women with gestational diabetes (GDM) and women without GDM suggest a possible alteration in fatty acid metabolism in GDM. Data from systematic reviews show a consistent association between marine or algae oil supplementation with higher length of gestation, improvement in maternal mood and neural development. Nonetheless, few interventions on diet and PA have focused on metabolic control in obese women and their impacts have not been consistent. Additionally, few intervention studies have explored the effect of n3LC-PUFAs supplementation on pregnant women in the incidence of GDM, with no studies conducted in obese pregnant women. Therefore, combining an n3LC-PUFAs supplementation with a lifestyle intervention could enhance the metabolic control of obese pregnant women. We propose to evaluate the effects of an n3LC-PUFAs supplementation intervention among obese pregnant women (independently and combined with a diet and physical activity intervention) on metabolic control in mothers and their offspring.

In 2013 we started in 12 primary health clinics (PHCC) of the South East area of Santiago Chile a cluster randomized trial -the Chilean Maternal & Infant Nutrition Cohort Study (CHiMINCs)- that aims to improve weight control during pregnancy and offspring growth during infancy by enhancing PHCC's maternal and infant weight monitoring systems as well as promoting breastfeeding. In the current study we propose to expand that effort trying to optimize metabolic control of obese pregnant women and their offspring by combining home-based diet and physical activity counseling and n3LC-PUFAs supplementation. Women who seek prenatal care in any of the 12 selected PHCC with <14 weeks gestation at first prenatal visit; body mass index (BMI) >30 Kg/m2 at first prenatal visit; have a singleton pregnancy will be asked to participate. We will recruit 1000 women; 250 women per arm of the study. After randomization, obese pregnant women in the intervention group 1 will receive home-based Diet & Physical activity (PA) counseling plus n3LC-PUFAs oral supplementation based on Schizochytrium oil (S-oil) containing 800 mg docosahexaenoic (DHA) acid/day, which will be administered as capsular preparations containing 200 mg DHA/capsule (4 capsules/day). Obese pregnant women in the intervention group 2 will receive the standard education sessions included in the prenatal controls at PHCC but no home-based counseling sessions, plus n3LC-PUFAs supplementation of 800 mg of DHA. Obese pregnant women in the intervention group 3 will receive the home-based diet & PA counseling sessions plus n3LC-PUFAs placebo that will consist of S-oil containing 200 mg DHA/day. Placebo will be administered as capsular preparations containing 50 mg DHA/capsule (4 capsules/day), given that evidence suggests that it would be unethical not to provide DHA during pregnancy. Placebo will be delivered in the same way that the n3LC-PUFA supplementation. The control group will receive routine diet & PA PHCC counseling sessions plus placebo (4 capsules of 50 mg DHA per day). Measurements will be collected at baseline (<14 weeks of pregnancy), mid-pregnancy (24-28 weeks), and at delivery. Baseline and 24-28 weeks measurements will be carried out at home.

Analyses will be done according both to the "intention-to-treat" (i.e. effectiveness approach) and "per protocol" (i.e. efficacy approach) principles. In accordance with the 2×2 factorial design, the diet & PA intervention (Intervention Groups 1 and 3) will be compared to the routine care intervention (Intervention Groups 2 and Control Group) and the n3LC-PUFAs supplementation intervention (Intervention Groups 1 and 2) will be compared to placebo (Intervention Group 3 and Control Group). To evaluate the effects of the two combined interventions the outcomes in each of the 3 intervened groups will be compared between them and with the outcomes in the control group. We expect that the intervention will contribute to achieving a better metabolic control during pregnancy. Ultimately, we expect that this study will contribute to advance the understanding of how to develop and implement effective actions to promote healthier pregnancies and therefore, healthier lives for mothers and their offsprings.

ELIGIBILITY:
Inclusion Criteria:

* ≤14 weeks gestational age at first prenatal visit
* Body mass index (BMI) >30 Kg/m2 at first prenatal visit
* Have a singleton pregnancy
* Plan to deliver at the "Sotero del Rio Hospital".

Exclusion Criteria:

* Preexisting diabetes (known or diagnosed at first control (Fasting Plasma Glucose > 126 mg/dl or 2h plasma glucose > 200 mg/dl during an oral glucose tolerance test (OTTG))
* Insulin or metformin use
* Known medical or obstetric complications which restrict physical activity
* History of eating disorders
* High risk for hemorrhagic bleeding
* High risk pregnancy according to national guidelines

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1002 (Actual)
Dates: Start 2015-08; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Gestational Diabetes Mellitus (GDM) | 24-28 weeks of gestation
  According to ADA 2011 guidelines (fasting glucose ≥92 mg/dL and/or 2 h after ≥153 mg/dL)
Macrosomia | At birth
  Birth weight greater than 4000 g
Prevalence of insulin resistance | At birth
  Prevalence of insulin resistance (IR) defined as cord blood homeostasis model assessment-estimated insulin resistance (HOMA-IR) > 2.60 at birth.

SECONDARY OUTCOMES:
Low Birth Weight | At birth
  Birth weight below 2500 g
Excess weight gain during pregnancy | Self reported pre-gestational weight, weight gain will be measured at least three times at 10-14, 24-28, 35-37 weeks of gestation, and also at delivery
  Weight at delivery minus the pregestational weight
Pre-eclampsia | 24-28 weeks of gestation
  Blood pressure ≥ 140 mm Hg systolic or ≥ 90 mm Hg diastolic
Preterm delivery | At birth
  Child´s birth < 37 weeks gestational age
Proportions of cesareans | At birth
  Proportion of children delivered via cesarean section divided total of deliveries

CONTACTS AND LOCATIONS:
Overall Officials: MARIA LUISA GARMENDIA, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Institute of Nutrition and Food Technology, Santiago, Chile

REFERENCES:
- [Derived] Garmendia ML, Casanello P, Flores M, Kusanovic JP, Uauy R. The effects of a combined intervention (docosahexaenoic acid supplementation and home-based dietary counseling) on metabolic control in obese and overweight pregnant women: the MIGHT study. Am J Obstet Gynecol. 2021 May;224(5):526.e1-526.e25. doi: 10.1016/j.ajog.2020.10.048. Epub 2020 Nov 2. PMID 33152314
- [Derived] Garmendia ML, Corvalan C, Casanello P, Araya M, Flores M, Bravo A, Kusanovic JP, Olmos P, Uauy R. Effectiveness on maternal and offspring metabolic control of a home-based dietary counseling intervention and DHA supplementation in obese/overweight pregnant women (MIGHT study): A randomized controlled trial-Study protocol. Contemp Clin Trials. 2018 Jul;70:35-40. doi: 10.1016/j.cct.2018.05.007. Epub 2018 May 17. PMID 29777864